CLINICAL TRIAL: NCT03646396
Title: Effect of Daclatasvir Plus Sofosbuvir on Angiogenesis in Egyptian Patients With Chronic HCV Infection
Brief Title: Effect of Sofosbuvir-daclatasuvir on Angiogenesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, PhDTropical Medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sofosbuvir angiogenesis
Record Dates: First submitted 2018-08-23; First posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: HCV Coinfection

STUDY DESIGN:
Intervention Model Description: Drug "sof-Dakla"
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sofosbuvir-daclatasvir (Experimental): Sofosbuvir-daclatasvir for 3 months
  Interventions: Drug: Sofosbuvir-daclatasvir

INTERVENTIONS:
Drug: Sofosbuvir-daclatasvir — Sofosbuvir-daclatasvir for 3 months
  Other Names: sof-dakla

SUMMARY:
The study aimed at study of the Effect of Daclatasvir Plus Sofosbuvir on Angiogenesis in Egyptian Patients With Chronic HCV Infection

DETAILED DESCRIPTION:
The study primary aim was at evaluation of the Effect of Daclatasvir Plus Sofosbuvir on Angiogenesis in Egyptian Patients With Chronic HCV Infection

ELIGIBILITY:
Inclusion Criteria:

* Chronic HCV patients

Exclusion Criteria:

* HCC.
* HIV or HBV.
* Malignancy.
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with change in VEGF, TGFB1 | 6 months
  Number of patients with change in VEGF, TGFB1

CONTACTS AND LOCATIONS:
Overall Officials: Eman h abd El-Razek, Msc, Principal Investigator — Clinical pharmacy Department- Tanta University; Tarek M Mostafa, Ph D, Principal Investigator — Clinical pharmacy Department- Tanta University; Nashwa Shebl, Ph D, Principal Investigator — Hematology and Gastroenterology - Menoufia University
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided